CLINICAL TRIAL: NCT01972113
Title: Vitamin K and Glucose Metabolism in Children at Risk for Diabetes
Brief Title: Vitamin K and Glucose Metabolism in Children at Risk for Diabetes (Vita-K 'n' Kids Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Collaborators: University of Alabama at Birmingham (Other); Yale University (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Norman Pollock, Associate Professor, Department of Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 611523 (Pro00000912); 16GRNT31090037 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Insulin Resistance; Insulin Sensitivity; Prediabetes; Dyslipidemia; Diabetes
Keywords: Vitamin K; Vitamin K2; Menaquinone-7; Osteocalcin; Children; Obesity; Insulin resistance; Insulin sensitivity; Beta-cell function; Prediabetes; Matrix Gla protein; Arterial stiffness; Endothelial function
MeSH Terms: conditions — Obesity; Insulin Resistance; Prediabetic State; Dyslipidemias; Diabetes Mellitus | interventions — Vitamin K 2; menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo-Control (Placebo Comparator): The placebo-control group will take one placebo softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: Placebo-Control
- Low-Dose Vitamin K2 (45 mcg/d) (Active Comparator): The low-dose vitamin K2 group will take one 45-mcg vitamin K2 softgel capsule and one placebo softgel capsule every day for 8 weeks.
  Interventions: Dietary Supplement: Low-Dose Vitamin K2 (menaquinone-7; 45 mcg/d)
- High-Dose Vitamin K2 (90 mcg/d) (Active Comparator): The high-dose vitamin K2 group will take one 90-mcg vitamin K2 softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: High-Dose Vitamin K2 (menaquinone-7; 90 mcg/d)

INTERVENTIONS:
Dietary Supplement: Placebo-Control — one placebo softgel capsules per day (for 8 weeks) containing no vitamin K2 (menaquinone-7)
  Arms: Placebo-Control
Dietary Supplement: Low-Dose Vitamin K2 (menaquinone-7; 45 mcg/d) — one 45-mcg vitamin K2 (menaquinone-7) softgel capsule per day and one placebo softgel per day (containing no menaquinone-7) for 8 weeks
  Other Names: menaquinone-7
  Arms: Low-Dose Vitamin K2 (45 mcg/d)
Dietary Supplement: High-Dose Vitamin K2 (menaquinone-7; 90 mcg/d) — one 90-mcg vitamin K2 (menaquinone-7) softgel capsules per day for 8 weeks
  Other Names: menaquinone-7
  Arms: High-Dose Vitamin K2 (90 mcg/d)

SUMMARY:
The undercarboxylated fractions of the two vitamin K-dependent proteins osteocalcin and matrix Gla protein have been shown to play key roles in type 2 diabetes and cardiovascular disease (at least in mouse models). Clinical trials are needed to isolate the effects of vitamin K manipulation on carboxylation of these two proteins (osteocalcin and matrix GLA protein) and their subsequent effects on markers of diabetes and cardiovascular disease risk. The purpose of this pilot randomized, double-blind, placebo-controlled trial in children is to estimate the effective dose of vitamin K2 (menaquinone-7) supplementation (to improve carboxylation of both osteocalcin and matrix Gla protein), and whether it can have an effect on markers associated with diabetes and cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 17 years
* BMI less than 85th percentile for age and gender
* Subject and parent/guardian understands the study protocol and agrees to comply with it
* Informed Consent Form signed by the parent/guardian and assent signed by the subject

Exclusion Criteria:

* Subjects using vitamin supplements containing vitamin k
* Subjects with (a history of) metabolic or gastrointestinal diseases including hepatic disorders
* Subjects presenting chronic degenerative and/or inflammatory diseases
* Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters (salicylates, antibiotics)
* Subjects receiving corticosteroid treatment
* Subjects using oral anticoagulants
* Subjects with a history of soy allergy
* Subjects who have participated in a clinical study more recently than one month before the current study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum lipid concentrations | 8 weeks
  To determine if vitamin K supplementation improves fasting lipid panel (triglycerides, total cholesterol, HDL-cholesterol, and LDL-cholesterol) in a dose-dependent manner.
Change in insulin sensitivity | 8 weeks
  To determine if vitamin K supplementation improves insulin sensitivity in a dose-dependent manner. Insulin sensitivity will be calculated from plasma insulin and glucose concentrations measured during a 2-hour glucose tolerance test by using the oral glucose minimal model.
Change in beta-cell function | 8 weeks
  To determine if vitamin K supplementation improves insulin sensitivity in a dose-dependent manner. Beta-cell function, as assessed by dynamic beta-cell responsitivity, will be calculated from plasma glucose and C-peptide concentrations measured during a 2-hour glucose tolerance test by using the oral C-peptide minimal model.

SECONDARY OUTCOMES:
Change in coagulation | 8 weeks
  Coagulation-related parameters (i.e., prothrombin time and activated partial thromboplastin time) will be assessed at baseline and 8 weeks to assess clotting function.
Change in arterial stiffness (pulse wave velocity) | 8 weeks
  Arterial stiffness, as measured by pulse wave velocity (PWV), will be assessed at baseline and 8 weeks to explore whether change in arterial stiffness is influenced by vitamin K2 supplementation.
Change in endothelial function (Flow-mediated dilation) | 8 weeks
  Endothelial function, as measured by flow-mediated dilation (FMD), will be assessed at baseline and 8 weeks to explore whether change in endothelial function is influenced by vitamin K2 supplementation.
Effects of sex, race, bone age, and pubertal stage on changes in glucosemetabolism (insulin sensitivity and beta-cell function) | 8 weeks
  Moderation effects of sex, race, bone age, and pubertal stage in the associations of vitamin K-induced changes in carboxylation of osteocalcin on markers of glucose metabolism will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Pollock, Ph.D., Principal Investigator — Department of Medicine, Medical College of Georgia, Augusta University
Locations (1):
- Medical College of Georgia; Augusta University, Augusta, Georgia, United States

REFERENCES:
- [Background] Pollock NK, Bernard PJ, Gower BA, Gundberg CM, Wenger K, Misra S, Bassali RW, Davis CL. Lower uncarboxylated osteocalcin concentrations in children with prediabetes is associated with beta-cell function. J Clin Endocrinol Metab. 2011 Jul;96(7):E1092-9. doi: 10.1210/jc.2010-2731. Epub 2011 Apr 20. PMID 21508147
- [Background] Gower BA, Pollock NK, Casazza K, Clemens TL, Goree LL, Granger WM. Associations of total and undercarboxylated osteocalcin with peripheral and hepatic insulin sensitivity and beta-cell function in overweight adults. J Clin Endocrinol Metab. 2013 Jul;98(7):E1173-80. doi: 10.1210/jc.2013-1203. Epub 2013 Apr 24. PMID 23616149
- [Background] Booth SL, Centi A, Smith SR, Gundberg C. The role of osteocalcin in human glucose metabolism: marker or mediator? Nat Rev Endocrinol. 2013 Jan;9(1):43-55. doi: 10.1038/nrendo.2012.201. Epub 2012 Nov 13. PMID 23147574
- [Background] Pollock NK. Childhood obesity, bone development, and cardiometabolic risk factors. Mol Cell Endocrinol. 2015 Jul 15;410:52-63. doi: 10.1016/j.mce.2015.03.016. Epub 2015 Mar 27. PMID 25817542
- [Background] Douthit MK, Fain ME, Nguyen JT, Williams CF, Jasti AH, Gutin B, Pollock NK. Phylloquinone Intake Is Associated with Cardiac Structure and Function in Adolescents. J Nutr. 2017 Oct 1;147(10):1960-1967. doi: 10.3945/jn.117.253666. PMID 28794209
- [Background] Fain ME, Kapuku GK, Paulson WD, Williams CF, Raed A, Dong Y, Knapen MHJ, Vermeer C, Pollock NK. Inactive Matrix Gla Protein, Arterial Stiffness, and Endothelial Function in African American Hemodialysis Patients. Am J Hypertens. 2018 May 7;31(6):735-741. doi: 10.1093/ajh/hpy049. PMID 29635270